CLINICAL TRIAL: NCT03924609
Title: Impact of Intensive Follow-up for Bone Metastasis on Characteristics and Prognosis of Chinese Breast Cancer Patients: A Multicenter Retrospective Study
Brief Title: Impact of Intensive Follow-up for Bone Metastasis on Characteristics and Prognosis of Chinese Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Fudan University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20160504
Record Dates: First submitted 2019-03-08; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Bone Metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone metastasis screening: The information about bone metastasis screening is retrospectively collected.
  Interventions: Diagnostic Test: Intensive screening / routine screening

INTERVENTIONS:
Diagnostic Test: Intensive screening / routine screening — Recommendation and results of bone imaging such as bone scan or PET/CT, or bone CT /MR are collected.

SUMMARY:
The purpose of this study is to retrospectively collect and analyse the characteristics of breast cancer patients with bone metastasis, and compare the impact of intensive follow-up with standard post-operative surveillance on survival of Chinese breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignant tumors in women, and the incidence rate is gradually increasing, accounts for the first place in the incidence of female malignant tumors. Bone metastasis is the most common distant metastatic site for breast cancer, accounting for approximately 70% of all patients with advanced breast cancer. About 26%-50% of breast cancer patients with primary metastases are bone. Autopsy results showed that the overall incidence of breast cancer bone metastasis was about 47%-85%.

Postoperative routine screening for bone metastases in breast cancer patients, whether domestic or foreign, is not recommended in most guidelines. These recommendations were based on two prospective randomized controlled trials in Italy in 1990s, indicated that a bone scan every six months or annually didn't provide a survival benefit to the patient. However, there were researches showing that about 11% of patients with asymptomatic breast cancer have bone metastases, suggesting that early screening might detect more patients with asymptomatic bone metastases. The meta-analysis also pointed out that early screening may prolong the disease-free survival of patients. Besides, the imaging techniques have advance rapidly and remarkably since then. New trials are needed to figure out whether imaging screening of asymptomatic patients should be routinely performed to detect more asymptomatic bone metastases needs further investigation.

ELIGIBILITY:
Inclusion Criteria:

A. Histologically proven breast cancer confirmed by biopsy or pathological examination of the resected tumor.

B. Histologically confirmed breast cancer patients, fulfilling any of the following:

1. . Multiple bone metastases indicated by bone scan
2. . Bone scan positive, and proven by other imaging examinations, including computed tomography (CT), magnetic resonance imaging (MRI) and X-ray.
3. . Bone scan positive, with clinical symptoms, including bone pain, pathologic fracture, spinal cord compression and so on.
4. . Bone metastases indicated by PET-CT
5. . Histologically proven bone metastases

Exclusion Criteria:

A. No bone metastases confirmed by pathological examination B. Bone metastases secondary to other malignant tumor other than breast cancer C. Secondary primary tumor

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 1500 breast cancer patients with bone metastasis diagnosed between 2006 and 2011
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 60 months, and bone scan is repeated every 12 months
  defined as the period from randomization to death from any cause, and it is censored at the last follow-up date when the patient is alive

SECONDARY OUTCOMES:
disease-free survival | 60 months, and bone scan is repeated every 12 months
  defined as time to disease recurrence (invasive local, regional, or distant metastasis) or death from any cause
distant metastasis-free survival | 60 months, and bone scan is repeated every 12 months
  defined as time to distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Rosselli Del Turco M, Palli D, Cariddi A, Ciatto S, Pacini P, Distante V. Intensive diagnostic follow-up after treatment of primary breast cancer. A randomized trial. National Research Council Project on Breast Cancer follow-up. JAMA. 1994 May 25;271(20):1593-7. doi: 10.1001/jama.271.20.1593. PMID 7848404
- [Background] Impact of follow-up testing on survival and health-related quality of life in breast cancer patients. A multicenter randomized controlled trial. The GIVIO Investigators. JAMA. 1994 May 25;271(20):1587-92. doi: 10.1001/jama.1994.03510440047031. PMID 8182811
- [Background] Palli D, Russo A, Saieva C, Ciatto S, Rosselli Del Turco M, Distante V, Pacini P. Intensive vs clinical follow-up after treatment of primary breast cancer: 10-year update of a randomized trial. National Research Council Project on Breast Cancer Follow-up. JAMA. 1999 May 5;281(17):1586. doi: 10.1001/jama.281.17.1586. No abstract available. PMID 10235147
- [Background] Rojas MP, Telaro E, Russo A, Moschetti I, Coe L, Fossati R, Palli D, del Roselli TM, Liberati A. Follow-up strategies for women treated for early breast cancer. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001768. doi: 10.1002/14651858.CD001768.pub2. PMID 15674884
- [Background] Gradishar WJ, Anderson BO, Balassanian R, Blair SL, Burstein HJ, Cyr A, Elias AD, Farrar WB, Forero A, Giordano SH, Goetz M, Goldstein LJ, Hudis CA, Isakoff SJ, Marcom PK, Mayer IA, McCormick B, Moran M, Patel SA, Pierce LJ, Reed EC, Salerno KE, Schwartzberg LS, Smith KL, Smith ML, Soliman H, Somlo G, Telli M, Ward JH, Shead DA, Kumar R. Invasive Breast Cancer Version 1.2016, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2016 Mar;14(3):324-54. doi: 10.6004/jnccn.2016.0037. PMID 26957618
- [Background] Khatcheressian JL, Hurley P, Bantug E, Esserman LJ, Grunfeld E, Halberg F, Hantel A, Henry NL, Muss HB, Smith TJ, Vogel VG, Wolff AC, Somerfield MR, Davidson NE; American Society of Clinical Oncology. Breast cancer follow-up and management after primary treatment: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2013 Mar 1;31(7):961-5. doi: 10.1200/JCO.2012.45.9859. Epub 2012 Nov 5. PMID 23129741
- [Background] Yong M, Jensen AO, Jacobsen JB, Norgaard M, Fryzek JP, Sorensen HT. Survival in breast cancer patients with bone metastases and skeletal-related events: a population-based cohort study in Denmark (1999-2007). Breast Cancer Res Treat. 2011 Sep;129(2):495-503. doi: 10.1007/s10549-011-1475-5. Epub 2011 Apr 2. PMID 21461730
- [Background] Gong Y, Liu YR, Ji P, Hu X, Shao ZM. Impact of molecular subtypes on metastatic breast cancer patients: a SEER population-based study. Sci Rep. 2017 Mar 27;7:45411. doi: 10.1038/srep45411. PMID 28345619
- [Background] Xiong Z, Deng G, Huang X, Li X, Xie X, Wang J, Shuang Z, Wang X. Bone metastasis pattern in initial metastatic breast cancer: a population-based study. Cancer Manag Res. 2018 Feb 9;10:287-295. doi: 10.2147/CMAR.S155524. eCollection 2018. PMID 29467583
- [Background] Zhang H, Zhu W, Biskup E, Yang W, Yang Z, Wang H, Qiu X, Zhang C, Hu G, Hu G. Incidence, risk factors and prognostic characteristics of bone metastases and skeletal-related events (SREs) in breast cancer patients: A systematic review of the real world data. J Bone Oncol. 2018 Feb 3;11:38-50. doi: 10.1016/j.jbo.2018.01.004. eCollection 2018 Jun. PMID 29511626
- [Background] Coleman R, de Boer R, Eidtmann H, Llombart A, Davidson N, Neven P, von Minckwitz G, Sleeboom HP, Forbes J, Barrios C, Frassoldati A, Campbell I, Paija O, Martin N, Modi A, Bundred N. Zoledronic acid (zoledronate) for postmenopausal women with early breast cancer receiving adjuvant letrozole (ZO-FAST study): final 60-month results. Ann Oncol. 2013 Feb;24(2):398-405. doi: 10.1093/annonc/mds277. Epub 2012 Oct 9. PMID 23047045